CLINICAL TRIAL: NCT06371885
Title: Shock Wave on Pillar Pain After Carpal Tunnel Release in Hand Burn
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Ahmed Elsayeh, Lecturer of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004646
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Hand Burn; Carpal Tunnel Syndrome
Keywords: Carpal Tunnel Syndrome; Hand Burn; Pillar pain; Shock wave therapy
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Interventional (clinical trial)
Who Masked: Participant
Masking Description: Double mask for both groups (participant)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shock wave therapy group (Active Comparator): This group will be composed of twenty-six patients who will managed by shock wave therapy one session per week, each ESWT session will involve 2,000 pulses of the focus probe at 4-bar pressure and 5 Hz frequency for twelve weeks in addition to the traditional physical therapy in form of (10 minutes hot pack around wrist and forearm and 10 minutes of gentle stretching exercises for wrist joint, three sessions per week for twelve weeks.
  Interventions: Device: shock wave therapy; Other: traditional physical therapy
- Control group (Active Comparator): This group will be composed of twenty-six patients who will only managed by the traditional physical therapy in form of (10 minutes hot pack around wrist and forearm and 10 minutes of gentle stretching exercises for wrist joint, three sessions per week for twelve weeks
  Interventions: Other: traditional physical therapy

INTERVENTIONS:
Device: shock wave therapy — shock wave therapy will be applied one session per week, each ESWT session will involve 2,000 pulses of the focus probe at 4-bar pressure and 5 Hz frequency for twelve weeks
  Arms: Shock wave therapy group
Other: traditional physical therapy — the traditional physical therapy will be in form of (10 minutes hot pack around wrist and forearm and 10 minutes of gentle stretching exercises for wrist joint, three sessions per week for twelve weeks

SUMMARY:
"In burn cases, the reported causes of CTS are increased volume of carpal tunnel content due to edema and synovitis, wrist hyperextension, tight dressing, fibrosis, and direct burn to the nerve. There are two types of pain that occur in the palm of the hand after carpal tunnel surgery: incisional pain and pillar pain. The incision pain typically only lasts for a few days or weeks after surgery, while the pillar pain occurs on the sides of the incision in the thicker parts of the palm, called the thenar and hypothenar eminences. This is where the transverse ligament attaches to the carpal bones, forming the carpal tunnel.

So, in this study we will find out if shock wave therapy has therapeutic effect on pillar pain after carpal tunnel release in hand burn.

DETAILED DESCRIPTION:
The development of CTS following burns is common and usually occurs due to thermal burns, owing to excessive edema in circumferential burns, extensive metabolic and inflammatory changes occur in response to burnCarpal tunnel release surgery is one of the most common procedures performed by hand surgeons. Pillar pain is a frequent symptom following carpal tunnel release. The pain is located at the base of the hand in the heel of the palm. The muscles at the thumb base (thenar eminence) and the muscles at the base of the small finger (hypothenar eminence) are the usual areas of tenderness. The palm is sore when pressed in these locations, marked with red asterisks in the photo.

Shock wave therapy is a physical therapy modality that involves the administration of high-intensity sound waves arising from sudden pressure changes to the body. Those changes result in strong waves that cause compression and tension leading to anesthesia of the nerve fibers through biochemical changes and reduced inflammation in the soft tissue. It is believed that the release of angiogenesis-related growth factors of the mechanism of action in the soft tissues after shock wave accelerates the formation of new vessels and increases oxygenation in the environment, resulting in accelerated tissue recovery.

So, in this study we will find out if shock wave therapy has therapeutic effect on pillar pain after carpal tunnel release in hand burn. In this single blind randomized clinical trial, Fifty- two patients who had upper limb burn with the percentage of the total body surface area ranging from 20 % to 25 % and diagnosed as a 2nd or 3rd degree burn complicated with carpal tunnel syndrome, their ages range between 20 and 35 years, will be recruited from the outpatient clinic of burn in Mansoura hospitals. The patients will be randomly assigned into two equal groups. Sock wave group and control group.

Shock wave therapy group:

This group will be composed of twenty-six patients who will managed by shock wave therapy one session per week, each ESWT session will involve 2,000 pulses of the focus probe at 4-bar pressure and 5 Hz frequency for twelve weeks in addition to the traditional physical therapy.

Control group:

This group will be composed of twenty-six patients who will only managed by the traditional physical therapying form of (10 minutes hot pack around wrist and forearm and 10 minutes of gentle stretching exercises for wrist joint, three sessions per week for twelve weeks.

The outcome measures will be assessed using Visual Analog Scale, Hand held dynamometer, and Michigan hand out Comes questionnaire before and after 12 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age range will be from 20 to 35 years.
* Patients who have upper limb burn with the percentage of the total body surface area ranging from 20 % to 25 % and diagnosed as a 2nd or 3rd degree burn and complicated with carpal tunnel syndrome post burn. The diagnosis will be confirmed by using electroneurographic (ENG) examination as well as by using physical examination which included Tinel's test and Phalen's test.
* All patients are non-smokers and are under own prescribed medications described by their physicians.

Exclusion Criteria:

* Sensory or motor neuropathy.
* Systemic inflammatory diseases.
* A history of surgery other than CTRS or trauma/fracture in the hand and hand-wrist region.
* Local infections at the hand level.
* Pregnancy.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Change from baseline at twelve weeks after the intervention
  It is a pain rating scale. Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm)
Hand held dynamometer | Change from baseline at twelve weeks after the intervention
  It is a test to measure the maximum isometric strength of the hand and forearm muscles. Handgrip strength is important for any sport in which the hands are used for catching, throwing or lifting.

SECONDARY OUTCOMES:
Michigan hand out Comes questionnaire | Change from baseline at twelve weeks after the intervention
  t is a tool used to assess patients with hand disorders through the measurement of 6 health domains: overall hand function, activities of daily living (ADLs), pain, work performance, aesthetics, and patient satisfaction. The MHQ is a 57-item patient-reported outcome measure in hand surgery. The scale assesses six domains: overall hand function, activities of daily living, pain, work performance, aesthetics, and satisfaction with hand function. Each item is scored on a scale of 1 to 5. A domain score ranges from 0 (worst) to 100 (best), with higher scores indicating better hand function. However, the total score of a "pain domain" is reversed ("0 = best" to "100 = worst"), and therefore, a higher score in that domain indicates greater pain.

CONTACTS AND LOCATIONS:
Overall Officials: Shaimaa MA El Sayeh, Study Director — Lecturer at Faculty of Physical Therapy, Cairo University
Locations (1):
- Shaimaa Mohamed Ahmed El Sayeh, Cairo, New Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No